CLINICAL TRIAL: NCT02502162
Title: Low-Dose Naltrexone for the Treatment of Complex Regional Pain Syndrome
Acronym: LDN-CRPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Sean Mackey, Redlich Professor Departments of Anesthesiology, Perioperative and Pain Medicine | Neurosciences | Neurology (by courtesy), Chief, Division of Pain Medicine, Director, Stanford Systems Neuroscience and Pain Lab (SNAPL), Stanford University, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 33607
Record Dates: First submitted 2015-07-15; First posted 2015-07-20 (Estimated); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Complex Regional Pain Syndrome
MeSH Terms: conditions — Complex Regional Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LDN (Experimental): Naltrexone HCL, 4.5 mg, Once a day.
  Interventions: Drug: LDN
- Placebo (Placebo Comparator): Sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LDN
  Arms: LDN
Drug: Placebo — Sugar pill
  Arms: Placebo

SUMMARY:
The investigators are testing treatment with low-dose naltrexone (LDN) for symptom relief of complex regional pain syndrome (CRPS). Study participants will be randomly assigned to receive either LDN or placebo for a period of several weeks. During this period participants will be asked to attend either in-person or virtual study visits and complete questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Upper and/or lower extremity CRPS
* On stable treatment for 1 month
* CRPS for at least 1 year
* Meet the Budapest criteria for CRPS at time of the study.

Exclusion Criteria:

* Any known allergy to naltrexone or naloxone
* Use of prescription opioid analgesics or illegal opioid use
* Current or planned pregnancy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-06; Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Changes in pain severity | Approximately 4 weeks after conclusion of treatment.
  Daily pain reports on a 0-10 numerical rating scale for pain, where 0=no pain and 10=pain as bad as you can imagine

CONTACTS AND LOCATIONS:
Overall Officials: Sean Mackey, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States